CLINICAL TRIAL: NCT00872846
Title: Evaluation of the BALANCE System in Type 2 Diabetic Patients
Brief Title: Balance System Study in Type 2 Diabetic Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Beta-Stim Ltd. (Industry)
Collaborators: Meditrial Europe Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 598500
Record Dates: First submitted 2009-03-28; First posted 2009-03-31 (Estimated); Last update posted 2012-01-24 (Estimated); Status verified 2012-01

CONDITIONS: Type 2 Diabetes; Obesity
Keywords: Body weight; Signs and symptoms; Obesity; Metabolic disease; Diabetes mellitus type 2; Diabetes mellitus; Nutrition disorder; Endocrine system diseases; Overweight; Overnutrition; Glucose metabolic disorder
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity; Body Weight; Signs and Symptoms; Metabolic Diseases; Diabetes Mellitus; Nutrition Disorders; Endocrine System Diseases; Overweight; Overnutrition; Glucose Metabolism Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: BALANCE System intestinal electrical stimulator — The BALANCE System stimulates the duodenum in a specialized way to strengthen the natural contractions and mimic the sensation of fullness (satiety). The patient is expected to feel full after eating smaller amounts of food than normal. In addition, duodenal stimulation has been shown to induce favorable changes in postprandial glucose levels, glucose tolerance testing and insulin levels.
  Other Names: BALANCE System

SUMMARY:
To evaluate the safety and performance of the BALANCE System in treating patients who have type 2 diabetes and are overweight. Impact on blood glucose levels, weight loss, blood pressure and other clinical and metabolic parameters will be studied.

DETAILED DESCRIPTION:
The BALANCE System stimulates the duodenum in a specialized way to strengthen the natural contractions and mimic the sensation of fullness (satiety). The patient is expected to feel full after eating smaller amounts of food than normal. In addition, duodenal stimulation has been shown to induce favorable changes in postprandial glucose levels, glucose tolerance testing and insulin levels.

The target population type II diabetic patients uncontrolled with oral medications, and with overweight (BMI >30). The Balance System may overcome the known disadvantages of insulin therapy and allow early treatment of these patients, potentially preventing the progression of obesity and diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 Diabetes inadequately controlled on a maximum of three oral anti-diabetic agents
* HbA1c between 7 and 10% inclusive
* Fasting Blood Glucose between 126 and 200 mg/dL
* Body Mass Index (BMI) in the range of 30.0 to 45.0 kg/m2
* Stable oral anti-diabetic therapy for at least 3 months
* Subjects who are able and willing to perform self monitoring of plasma glucose for the entire trial period
* Able and willing to sign informed consent and return for follow-up assessments

Exclusion Criteria:

* Type 1 Diabetes
* Subjects at high risk of general anesthesia or surgery
* Subjects with prior pancreatitis
* Subjects treated with insulin within three months of screening
* Female with a positive pregnancy test, planning to become pregnant during screening, active treatment, or the follow up period, breastfeeding, or judged to be using inadequate contraceptive methods.
* Subjects who underwent previous intra abdominal, GI tract surgery or a major abdominal trauma.
* Subjects with other implanted electrical stimulation devices
* Subjects with motility disorders of the GI tract such as gastroparesis
* Subjects who are receiving medications known to affect gastric motility
* Subjects with history of peptic ulcer disease
* Subjects with any serious health condition, such as cancer, cardiac diseases, immunodeficiency disorders, liver disease, pulmonary disease, renal insufficiency, coagulopathy or a major depressive disorder.
* Subjects with severe diabetic complications, such as retinopathy or nephropathy
* Subjects with metabolic or endocrine disorders like primary or secondary Cushing syndrome
* Subjects who received another investigational agent within 30 days prior to screening
* Evidence of current or recent alcohol or drug abuse within the past year prior to screening
* Subjects who are unlikely to be available for follow-up as specified in the protocol
* Subjects with a past or present psychiatric condition that may impair his or her ability to comply with the study procedures
* Subjects with history of volvulus
* Subjects with history of known small bowel adhesions or any known GI adhesions
* Subjects with deficiencies of known vitamins, e.g. B12
* Subjects with known celiac disease or inflammatory bowel disease
* Subjects with conditions that, in the judgment of the investigator, precludes successful participation to the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2009-02; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Evaluation of the of device and/or procedure related adverse events | 12 months

SECONDARY OUTCOMES:
Significant decrease in the HbA1c values from baseline | at week 4, and at month 2,3,4,5,6,8,10,12

CONTACTS AND LOCATIONS:
Overall Officials: Jakob R Izbicki, Prof. Dr. med, Principal Investigator — The University Medical Center Hamburg-Eppendorf (UKE), Department of General, Visceral- and Thoracic-Surgery, Germany
Locations (1):
- University Clinic Hamburg-Eppendorf (UKE), Hamburg, Germany